CLINICAL TRIAL: NCT01265719
Title: A Prospective, Non-interventional, Longitudinal Cohort Study To Evaluate The Long-term Safety Of Latanoprost Treatment In Pediatric Populations
Brief Title: Long-Term Non-Interventional Latanoprost Study
Acronym: LYNX
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111143; PFI-LAT-2009-01 (Other: Alias Study Number); LYNX (Other: Other identifier)
Record Dates: First submitted 2010-12-16; First posted 2010-12-23 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2018-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Prospective; non-interventional; longitudinal; cohort study
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Latanoprost-treatment group
  Interventions: Other: No intervention other than routine medical care
- Non-topical prostaglandin analogue treatment group
  Interventions: Other: No intervention other than routine medical care

INTERVENTIONS:
Other: No intervention other than routine medical care — Subjects continuously treated with Latanoprost for at least one month Latanoprost treatment during the study period.
  Other Names: Observational
  Groups: Latanoprost-treatment group
Other: No intervention other than routine medical care — Subjects not treated with any topical prostaglandin analogues or continuously treated with topical prostaglandin analogues for less than one month before the baseline examination, and unlikely to be treated with topical prostaglandin analogues during the study period.
  Other Names: Observational
  Groups: Non-topical prostaglandin analogue treatment group

SUMMARY:
This is a non-interventional, prospective, longitudinal cohort study. A total of 150 pediatric subjects with glaucoma or elevated intraocular pressure, including 75 latanoprost-treated subjects and 75 non-topical prostaglandin analogue treated subjects, will be enrolled from ophthalmic hospital clinics and academic ophthalmic centers. As a non-interventional study, the study subjects' continued use of latanoprost and assessments of ocular events will be obtained through the routine medical follow-up with treating ophthalmologists or other designated members of the medical care team.

DETAILED DESCRIPTION:
At least 40 subjects in each of the following age groups: 1-<5 years and 5-<18 years. No minimum required numbers in the <1 year age group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female <18 years of age (neonates must be at least 36 weeks gestational age).
* Diagnosis of pediatric glaucoma or elevated intraocular pressure.
* Evidence of a personally signed and dated informed consent document indicating that the subject (and/or a legally acceptable representative) has been informed of all pertinent aspects of the study. A signed and dated assent will be required where applicable according to local laws.

For treated subjects only:

* Continuously treated with latanoprost for at least 1 month within the year prior to the baseline examination.

For untreated subjects only:

* Continuously treated with latanoprost or other topical prostaglandin analogues for less than one month prior to the baseline examination (based on the best knowledge of treating ophthalmologists), and unlikely to be treated with latanoprost or other topical prostaglandin analogues during the three-year study period; OR
* No prior treatment with latanoprost or other topical prostaglandin analogues, and unlikely to be treated with latanoprost or other topical prostaglandin analogues during the three-year study period.

Exclusion Criteria:

* Unable/unwilling to comply with protocol.
* Pregnant or nursing females at baseline.
* For treated subjects only: a history of allergy or hypersensitivity to any of the ingredients contained in latanoprost (e.g., hypersensitivity to benzalkonium chloride).

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric populations diagnosed with glaucoma or elevated intraocular pressure
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Dienst Oftalmologie, Edegem
  - Universitair Ziekenhuis Leuven - Campus Sint-Raphaël, Leuven
- Clinica de Oftalmologia San Diego, Medellín, Antioquia, Colombia
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- Rigshospitalet - Glostrup, Glostrup Municipality, Denmark
- France (3):
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris, Cedex 19
  - CHU d'Amiens -Centre Saint Victor, Amiens
  - Hopital Claude Huriez, Lille
- Germany (3):
  - Universitaetsklinikum Giessen und Marburg, Giessen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Mainz, Mainz
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Greece
- Italy (4):
  - Azienda Ospedaliero Univ., Catania, CT
  - Ospedale Pediatrico Bambino Gesu, Fiumicino (Roma)
  - Istituto Giannina Gaslini, Divisione di Oculistica, Genova
  - Unita' Operativa di Oculistica Pediatrica, Azienda Ospedaliera Ospedale Niguarda Ca'Grande, Milan
- Óptima Visión, Miraflores, Lima region, Peru
- AIBILI - Associação para a Investigação Biomédica e Inovação em Luz e Imagem, Coimbra, Portugal
- Detska Fakultna nemocnica s poliklinikou Bratislava, Bratislava, Slovakia
- Spain (4):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Akademiska Sjukhuset, Uppsala
  - Ögonkliniken, Centrallasarettet, Västerås
- United Kingdom (3):
  - Manchester Royal Eye Hospital, Manchester, GT MAN
  - Birmingham and Midland Eye Centre, Consultant Ophthalmologist, Birmingham
  - Richard Desmond Childrens Eye Centre, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111143&StudyName=Long-Term%20Non-Interventional%20Latanoprost%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 175 patients were enrolled into the study in 14 countries in Europe and South America: 102 in the latanoprost treatment group and 73 in the non-Prostaglandin (PG) treatment group.
Pre-assignment Details: No significant events prior to group assignment are to be reported. This was a non-interventional, prospective, longitudinal cohort study. Pediatric patients with glaucoma or elevated intra ocular pressure (IOP) were enrolled into 2 groups: Latanoprost-treated patients and non-PG treated patients.
Groups:
- Latanoprost Group: Patients continuously treated with latanoprost for at least 1 month within 1 year before the baseline examination and treated with latanoprost during the study period.
  Patients continuously treated with latanoprost for at least 1 month within 1 year before the baseline examination only.
- Non Prostaglandin Group: Patients continuously treated with latanoprost or other topical PG analogues for less than 1 month before the baseline examination, and unlikely to be treated with latanoprost or other topical PG analogues during the study period.
  Patients not treated with latanoprost or other topical PG analogues before the baseline examination, and unlikely to be treated with latanoprost or other topical PG analogues during the study period.
Period: Overall Study
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Started | 102 | 73
Completed | 88 | 60
Not Completed | 14 | 13
Not completed — Does not meet entrance criteria | 0 | 3
Not completed — Other reasons | 2 | 0
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Lost to Follow-up | 2 | 7
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Latanoprost Group | Non Prostaglandin Group | Total
Number analyzed (Participants) | 102 | 73 | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.8 (4.96) | 6.4 (4.76) | 7.8 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 28 | 76
  Male | 54 | 45 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last Available Observation in Best Corrected Visual Acuity (BCVA) (Snellen or Equivalent)
Description: Patients familiar with the letters of the alphabet were evaluated using Snellen visual acuity. Patients who were unable or unfamiliar with the letters of the alphabet were evaluated using charts made up of numbers, pictures (eg, Schering's Children's Eye Chart or Allen Cards), E's, or Landolt's broken rings, and other methods which were equivalent to Snellen acuity eg, HOTV testing).
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Least Squares Mean (Standard Error); unit: logMar
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
logMar
  <5 years: number analyzed (Participants) | 4 | 16
  <5 years | 0.25 (0.17) | -0.07 (0.09)
  5 to <18 years: number analyzed (Participants) | 69 | 36
  5 to <18 years | 0.01 (0.02) | 0.04 (0.04)
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; <5 years; Test type: Superiority or Other; p = 0.1126, ANCOVA; LS Mean difference = 0.33, 95% CI 2-sided [-0.09 to 0.74], Standard Error of Mean 0.20 — Change from baseline to last available observation in BCVA was analyzed using an ANCOVA model with fixed effect for treatment group with baseline BCVA value as covariate
Statistical Analysis 2: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years; Test type: Superiority or Other; p = 0.4840, ANCOVA; LS Mean difference = -0.03, 95% CI 2-sided [-0.12 to 0.06], Standard Error of Mean 0.04 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Clinically Meaningful Change in Refractive Error
Description: The refractive error [cycloplegic where appropriate (eg, those unable to cooperate with manifest refraction)] were determined at the baseline visit and assessed at the following visits.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 8 | 2

3. Secondary Outcome: Change From Baseline to Last Available Observation in Horizontal Corneal Diameter (by Caliper and/or Ruler)
Description: The horizontal corneal diameter was measured along the horizontal meridians. Diameter was measured using either a series of transparent plates with holes of different diameters in quarter-millimeter increments or with calibrated calipers compared against a ruler. When using calipers, the corneal diameter measurement was taken from limbus to a similar point 180° away at the opposite limbus. When not examining the children with anesthesia, it was recommended to use a tape measure across the head while measuring horizontal corneal diameter by photographic method.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
mm
  <5 years: number analyzed (Participants) | 21 | 29
  <5 years | 0.33 (0.22) | 0.37 (0.19)
  5 to <18 years: number analyzed (Participants) | 68 | 36
  5 to <18 years | 0.08 (0.12) | 0.05 (0.16)
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; <5 years; Test type: Superiority or Other; p = 0.9020, ANCOVA; LS Mean difference = -0.04, 95% CI 2-sided [-0.63 to 0.56], Standard Error of Mean 0.30 — Change from baseline to last available observation in HCD was analyzed using an ANCOVA model with fixed effect for treatment group with baseline HCD value as covariate
Statistical Analysis 2: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years; Test type: Superiority or Other; p = 0.8826, ANCOVA; LS Mean difference = 0.03, 95% CI 2-sided [-0.37 to 0.43], Standard Error of Mean 0.20 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline to Last Available Observation in Intraocular Pressure (IOP)
Description: IOP was preferably measured using 1 of 3 applanation-contact methods: Goldmann applanation tonometry, Perkins tonometry, or TonoPen® (tonometry). iCare® rebound tonometer was also allowed if it was used consistently throughout the study.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
mmHg
  <5 years: number analyzed (Participants) | 21 | 30
  <5 years | -1.01 (0.94) | 0.61 (0.78)
  5 to <18 years, IOP <21mmHg at Baseline: number analyzed (Participants) | 65 | 33
  5 to <18 years, IOP <21mmHg at Baseline | 1.52 (0.43) | 1.62 (0.61)
  5 to <18 years, IOP ≥21mmHg at Baseline: number analyzed (Participants) | 10 | 4
  5 to <18 years, IOP ≥21mmHg at Baseline | -4.26 (1.22) | 2.40 (1.99)
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; <5 years; Test type: Superiority or Other; p = 0.2003, ANCOVA; LS Mean difference = -1.62, 95% CI 2-sided [-4.13 to 0.89], Standard Error of Mean 1.25 — Change from baseline to last available observation in IOP was analyzed using an ANCOVA model with fixed effect for treatment group with baseline IOP value as covariate
Statistical Analysis 2: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years (IOP <21mmHg at Baseline); Test type: Superiority or Other; p = 0.8940, ANCOVA; LS Mean difference = -0.10, 95% CI 2-sided [-1.59 to 1.39], Standard Error of Mean 0.75 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years (IOP ≥21mmHg at Baseline); Test type: Superiority or Other; p = 0.0184, ANCOVA; The results were interpreted with caution because of the very small sample size of non-PG treatment group (n=4); LS Mean difference = -6.66, 95% CI 2-sided [-11.95 to -1.36], Standard Error of Mean 2.41 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Cup-to-disc Ratio (for Assessment of Optic Nerve Changes/Structures) - Number of Participants With Clinically Significant Deterioration in Cup/Disc Ratios
Description: The cup/disc ratio was recorded horizontally and vertically for each examination, and reported in 0.1 increments.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 1 [-0.11 to 0.62] | 0
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; Test type: Superiority or Other; p > 0.999, Fisher Exact; Difference in percentage = 1.0, 95% CI 2-sided [-13.97 to 15.90]

6. Secondary Outcome: Visual Field Defects - Number of Participants With Clinically Significant Deterioration of Visual Field Defects.
Description: A visual field examination was performed for those patients who can cooperate automated perimetry utilizing a threshold program. All visual fields was conducted utilizing the standard white background with a Goldmann size III white stimulus. For those patients who can not perform formal visual field testing, then field to confrontation test was used for younger, non-verbal children, central, steady and maintains fixation was used.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 1 [-0.11 to 0.62] | 1
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; Test type: Superiority or Other; p > 0.999, Fisher Exact; Difference in percentage = -0.4, 95% CI 2-sided [-15.32 to 14.55]

7. Secondary Outcome: Iris Color Darkening
Description: Changes from baseline in iris color were reported at each follow-up visit. Photographs were taken at the discretion of investigators as per standard of care.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 4 [-0.11 to 0.62] | 2
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; Test type: Superiority or Other; p > 0.999, Fisher Exact; Difference in percentage = 1.2, 95% CI 2-sided [-13.78 to 16.09]

8. Secondary Outcome: Localized Pigmentation (Nevi or Freckles) of Conjunctiva, Iris and Choroid
Description: Changes from baseline in localized pigmentation (nevi and freckles) of the conjunctiva, iris and choroid were reported at each follow-up visit. Photographs were taken at the discretion of investigators as per standard of care.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 3 (0.17) [-0.11 to 0.62] | 3 (0.09)

9. Secondary Outcome: Eyelash Darkening/Thickening
Description: Changes from baseline in eyelash darkening/thickening/lengthening were reported at each follow-up visit. Photographs were taken at the discretion of investigators as per standard of care.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 3 [-0.11 to 0.62] | 1
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; Test type: Superiority or Other; p = 0.6414, Fisher Exact; Difference in percentage = 1.6, 95% CI 2-sided [-13.39 to 16.48]

10. Secondary Outcome: Change From Baseline to Last Available Observation in Length of Eyelash (by Caliper and/or Ruler)
Description: The longest eyelash (mm) measured by caliper or ruler was recorded at baseline and each follow-up visit.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
mm
  <5 years: number analyzed (Participants) | 19 | 28
  <5 years | 1.14 (0.40) | 0.53 (0.33)
  5 to <18 years: number analyzed (Participants) | 69 | 35
  5 to <18 years | 0.44 (0.19) | 0.65 (0.26)
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; <5 years; Test type: Superiority or Other; p = 0.2437, ANCOVA; LS Mean difference = 0.61, 95% CI 2-sided [-0.43 to 1.65], Standard Error of Mean 0.52 — Change from baseline to last available observation in longest lash length (LLL) was analyzed using an ANCOVA model with fixed effect for treatment group with baseline LLL value as covariate
Statistical Analysis 2: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years; Test type: Superiority or Other; p = 0.5199, ANCOVA; LS Mean difference = -0.21, 95% CI 2-sided [-0.85 to 0.43], Standard Error of Mean 0.32 — Change from baseline to last available observation in LLL was analyzed using an ANCOVA model with fixed effect for treatment group with baseline LLL value as covariate

11. Secondary Outcome: Change From Baseline to Last Available Observation in Corneal Thickness (Pachymeter)
Description: Central corneal thickness was measured using a calibrated pachymeter, preferably an ultrasonic pachymeter.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Least Squares Mean (Standard Error); unit: Micrometer
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Micrometer
  <5 years: number analyzed (Participants) | 16 | 21
  <5 years | -8.67 (11.51) | -5.99 (10.27)
  5 to <18 years: number analyzed (Participants) | 70 | 33
  5 to <18 years | 5.30 (2.75) | 6.17 (4.01)
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; <5 years; Test type: Superiority or Other; p = 0.8643, ANCOVA; LS Mean difference = -2.68, 95% CI 2-sided [-34.30 to 28.94], Standard Error of Mean 15.54 — Change from baseline to last available observation in corneal thickness was analyzed using an ANCOVA model with fixed effect for treatment group with baseline corneal thickness value as covariate
Statistical Analysis 2: Comparison: Latanoprost Group vs Non Prostaglandin Group; 5 to <18 years; Test type: Superiority or Other; p = 0.8591, ANCOVA; LS Mean difference = -0.87, 95% CI 2-sided [-10.54 to 8.80], Standard Error of Mean 4.87 — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Conjunctival/Ocular Hyperemia
Description: Conjunctiva hyperemia was assessed by slit-lamp examination. When slit-lamp examination is not possible due to subject cooperation, a fixation light and 20-diopter lens (for magnification) was used to assess this parameter. Conjunctival hyperemia was assessed and graded by ophthalmologist at baseline and follow-up visits from grades 0-3 and is as follows:
  0 = None, Normal: few vessels of palpebral or bulbar conjunctiva easily observed
  1. = Mild, Reddening of the palpebral or bulbar conjunctiva
  2. = Moderate, Bright reddening of the palpebral or bulbar conjunctiva
  3. = Severe, Deep, bright, and diffuse reddening of the palpebral or bulbar conjunctiva
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 6 [-0.11 to 0.62] | 1
Statistical Analysis 1: Comparison: Latanoprost Group vs Non Prostaglandin Group; Test type: Superiority or Other; p = 0.2413, Fisher Exact; Difference in percentage = 4.5, 95% CI 2-sided [-10.49 to 19.36]

13. Secondary Outcome: Number of Participants With a Change in Anterior Segment Biomicroscopy
Description: Slit-lamp biomicroscopy (mounted or hand-held) without fluorescein and without dilation of the pupil was performed. When slit-lamp examination was not possible, a fixation light and 20-diopter lens (for magnification) was used. At each scheduled visit, deposition of pigment on the corneal endothelial layer or the lens capsule or any abnormalities of the lids, conjunctivae, cornea, anterior chamber, iris, or lens was examined.
Time Frame: Evaluated at Baseline, 6 months, 12 months, 24 months and 36 months
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants | 0 (0.17) [-0.11 to 0.62] | 0 (0.09)

14. Secondary Outcome: Number of Participants With Abnormalities in Fundoscopy Posterior Segment at Baseline
Description: Fundoscopy was performed after dilation of the pupils (eg, 1 % tropicamide or cyclopentolate and 2 ½ % phenylephrine, or a clinically- appropriate dose according to the clinician's standard care of each particular patient). The examination included an evaluation of the vitreous body, retina (including the macula), and optic nerve head.
  The fundoscopy e-CRF was completed only at baseline because the investigators were required to perform slit lamp, direct or indirect ophthalmoscopy at each visit and report any AEs observed which included the vitreous, retina and optic nerve.
Time Frame: Evaluated at Baseline
Population: The Full Analysis population included all enrolled subjects.
Measure: Number; unit: Participants
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Number analyzed (Participants) | 102 | 73
Participants
  Vitreous body | 3 | 1
  Optic nerve head | 43 | 29
  Retina macula choroid | 12 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent throughout the entire study period or 28 calendar days after the last administration of latanoprost within the observational period, whichever is latest.
Description: One patient was missed in the adverse event raw data; no collection AE start date on case report form page hence the number of participants in Non Prostaglandin group is 72.
Arm/Group | Latanoprost Group | Non Prostaglandin Group
Serious Adverse Events (participants affected / at risk) | 11/102 | 2/72
Other Adverse Events (participants affected / at risk) | 20/102 | 14/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprost Group (N=102) | Non Prostaglandin Group (N=72)
Developmental glaucoma (Congenital, familial and genetic disorders) | 1 | 0
Neurofibromatosis (Congenital, familial and genetic disorders) | 1 | 0
Glaucoma (Eye disorders) | 2 | 0
Iris incarceration (Eye disorders) | 1 | 0
Posterior capsule opacification (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Intraocular pressure increased (Investigations) | 3 | 1
Optic nerve cup/disc ratio increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Eye operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprost Group (N=102) | Non Prostaglandin Group (N=72)
Conjunctival hyperaemia (Eye disorders) | 5 | 1
Eye pain (Eye disorders) | 4 | 0
Iris hyperpigmentation (Eye disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4
Intraocular pressure increased (Investigations) | 9 | 9

LIMITATIONS AND CAVEATS:
Inherent limitations of an observational study design (eg, lack of randomization), this was subject to the design/data-related limitations mainly Visual acuity, IOP, and visual field assessments in <5 years old age group were less reliable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.